CLINICAL TRIAL: NCT05185661
Title: Anemia Prevalence, Associated Factors, and Impact of eHealth Education Among School-going Adolescent Girls in Rural Bangladesh
Brief Title: Impact of eHealth Education to Reduce Anemia Among School-going Adolescent Girls in Rural Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: North South University, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Md Jiaur Rahman, PhD Researcher, Graduate School of Biomedical and Health Sciences, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021/OR-NSU/IRB/1102
Record Dates: First submitted 2021-12-04; First posted 2022-01-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anemia
Keywords: eHealth education; Anemia; Adolescents girl; Bangladesh
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Randomized control trial (RCT) study.
Masking Description: One school will be considered as an intervention group and another school control group to reduce the health education information bias between the intervention and control group participants through the coin toss simple randomization technique. Then computer-generated simple random sampling technique will be used to select anemic study participants for both the intervention and control group from the schools
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Two surveys: Demographic, lifestyle, hygiene-related (1) & knowledge, attitude, and practice (2) regarding anemia at baseline and end line of study.
  2. Investigations and physical examination will perform for CBC blood test except ESR, urine R/E, stool R/E, Height, weight for BMI, waist circumference, hip circumference, hip - waist ratio, and mid-upper arm circumference (MUAC) at baseline, mid-line, and end-line of study.
  Interventions: Behavioral: eHealth education
- Control Group (No Intervention): 1. Two surveys: Demographic, lifestyle, hygiene-related (1) & knowledge, attitude, and practice (2) regarding anemia at baseline and end line of study.
  2. Investigations and physical examination will perform for CBC blood test except ESR, urine R/E, stool R/E, Height, weight for BMI, waist circumference, hip circumference, hip - waist ratio, and mid-upper arm circumference (MUAC) at baseline, mid-line, and end-line of study.

INTERVENTIONS:
Behavioral: eHealth education — eHealth education intervention regarding the dietary plan, healthy-lifestyle, and hygiene:
  1. Group-wise eHealth education through online PowerPoint presentation session among study participants with their guardian: Two times (Before starting the intervention and mid-line; end of 4th-month intervention)
  2. eHealth education through phone calls & SMS
     * 1st to 4th month: 4 times in a month
     * 5th to 6th month: 3 times in a month
     * 6th to 8th month: 2 times in a month
  3. Control group will not get care and education
  Arms: Intervention Group

SUMMARY:
Adolescent girls are the highly vulnerable group to develop anemia due to reproductive immaturities, poor personal hygiene, lack of nutritional intake, and lack of health education in the rural area of Bangladesh. Rapid advantage of technology, eHealth is the promising tool to overcome the barriers and provide appropriate health guidelines in distant rural communities by developing knowledge, attitude, and practice to reduce anemia and mitigate risk among the school-going adolescent girls. This research aims (1) To evaluate eHealth education's impact on reducing anemia among adolescent girls in rural Bangladesh. (2) To assess the effect of eHealth education to change the knowledge, attitude, and practice among adolescent girls regarding anemia. A Randomized Control Trial study will be conducted from May 22, 2022, to January 21, 2023, in the two schools at the Chandpur district, Bangladesh. During the 8th months' intervention, will be provided eHealth education by the trained community health worker. The participant will be allocated who will be diagnosed as anemic through the blood hemoglobin screening. The sample size was calculated, and the total sample is 138. In this study, one school will be considered an intervention group and another school control group through the simple coin toss randomization technique. Then random sampling technique will be used to select study participants.

DETAILED DESCRIPTION:
Globally 1.62 billion people affect anemia, a significant public health threat, especially in low and middle-income countries (LMICs). The prevalence of anemia among non-pregnant and school-going is 30% and 25%, respectively, and 35% of this anemia in the LMICs. Anemia is a medical condition that can develop at any life stage, but at the reproductive age of women, adolescent girls (10-19 years), and growing children are susceptible. Adolescent age is a critical period of developmental transmission and reproductive maturation, requiring increased nutritional intake and proper health education; otherwise, it leads adolescents more vulnerable to future development. The primary reasons for developing anemia are the lack of iron-containing food intake, contaminated water, and poor sanitation. Also, the infection with soil-transmitted helminth is one of the leading blood losses causes of anemia.

Bangladesh is a middle-income, highly populated developing country. As per World Health Organization (WHO) 2019 data, Bangladesh has a 36.7% anemia prevalence among women of reproductive age. According to the WHO, if anemia prevalence is more than 40%, it is an alarming and severe public health problem. The whole-population anemia prevalence satisfies the criteria apparently; however, focusing on sub-population, it does not. For example, among the non-pregnant women's anemia, 73% live in rural Bangladesh. A scientific article reported that 51.6% of adolescent girls were suffering from anemia; 46%, 5.4%, and 0.2% were mild, moderate, severe anemia, respectively. Due to the high prevalence of rural women and adolescent girls' anemia in Bangladesh, adolescents are the highly venerable and more focused group. The lack of education, shortage of iron intake, poor economic status, poor personal hygiene, unhygienic toilets, parasitic infection are the main risk factors of anemia in Bangladesh. Proper interventions, including health education, should be provided to those vulnerable populations. i.e., adolescent girls in rural areas.

Lifestyle and behavioral change depend on knowledge, and nutritional knowledge is essential for good dietary habits. Health education is an effective way to increase knowledge. A school-based nutritional education reported that it is a feasible tool improving the hemoglobin level, knowledge, attitudes, and practices among adolescents. Health education is a useful approach to creating awareness among adolescent girls to reduce preventable diseases like anemia and build a future healthy mother.

In Bangladesh, mobile phone (85%) and network (99%) coverage are high among the rural communities, which is effective in delivering health education through eHealth technology. eHealth is the cost-effective and secure use of information and communications technologies supporting health and health-related fields, including health-care services, health surveillance, health literature, and health education, knowledge, and research (WHO E-Health Resolution 2005). mHealth is an important part of eHealth, which is the use of mobile and wireless technologies to support the achievement of health objectives and is viewed as having the potential to transform the face of health service delivery.

To investigators' knowledge, specific research is lacking about the effect of eHealth education among adolescent girls to create awareness and knowledge about the preventive, control, and risk reduction strategies of anemia in the school-going adolescent girls of rural Bangladesh. Moreover, knowledge gaps still exist regarding food habits and dietary practice, hygiene maintenance, lifestyle and behavior, medication adherence, etc., which are important factors developing anemia.

Knowledge gap:

To investigators' knowledge, specific research is lacking about the effect of eHealth education among adolescent girls to create awareness and knowledge about the preventive, control, and risk reduction strategies of anemia in the school-going adolescent girls of rural Bangladesh. Moreover, knowledge gaps still exist regarding food habits and dietary practice, hygiene maintenance, lifestyle and behavior, medication adherence, etc., which are important factors developing anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Who is diagnosed with mild and moderate anemia in the baseline screening of the study.
2. Who gives written consent to participate in the study through the legal guardian/participants.
3. Who is living and studying Chandpur district with assigned school for the study.

Exclusion Criteria:

1. Participants whose guardians/participants do not have a mobile phone will be excluded from the study.
2. Who is pregnant will be excluded from our study.
3. Who are physically and mentally sick will be excluded from our study.

3. Disagree to participate in this study

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The adolescent girl whose age is 10-19 years.
Enrollment: 138 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Impact of eHealth education to change the anemia level among school-going adolescent girls in rural areas of Bangladesh | 8 months after intervention
  Individuals school-going adolescent girls will be measured anemia level (No anemic, mild, moderate, and severe anemia) through the blood hemoglobin screening by the auto-hematology analyzer. According to WHO, 10-11 years adolescent girls Hb <11.5g/dl will be considered anemic, and <10-11.4, 7.0-9.9 g/dl, <7.0 g/dl will be considered mild, moderate, and severe anemia, respectively. Non-pregnant adolescent girls (12-19 years) Hb level < 12 g/dl will be considered suffering any form of anemia, and 10.0-11.9 g/dl, 7.0-9.9 g/dl, and <7.0 g/dl will be considered mild, moderate, and severe anemia, respectively. After eHealth education intervention, changes will be assessed (e.g., anemic to non-anemic, severe to mild/ moderate/non-anemic, moderate to mild/non-anemic, mild to non-anemic) from the baseline of anemia level among the school-going adolescent girls.

SECONDARY OUTCOMES:
Changes of knowledge, attitude, and practice regarding anemia among the school-going adolescent girls in rural areas of Bangladesh | 8 months after intervention
  The impact of eHealth education in changing knowledge, attitude, and practice regarding anemia will be assessed among school-going adolescent girls. Knowledge, attitude, and practice (KAP) will be measured through an adapted KAP model questionnaire of the Food and Agriculture Organization (FAO) at baseline and end of eight months of study. The questionnaire consisted of the multiple-choice options 'Yes', 'No,' and 'I don't know'. Correct responses will be given a score of 1, and incorrect responses will be given a score of 0. The option 'I don't know' will be considered as lack of knowledge and given a score of 0. KAP scores will be calculated by adding the number of correct answers divided by the total number of questions and multiplying by 100 to obtain a percentage score.

CONTACTS AND LOCATIONS:
Locations (1):
- Baburhat high school and Zubaida girl school, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jalambo M, Karim N, Naser I, Sharif R. Effects of iron supplementation and nutrition education on haemoglobin, ferritin and oxidative stress in iron-deficient female adolescents in Palestine: randomized control trial. East Mediterr Health J. 2018 Jul 29;24(6):560-568. doi: 10.26719/2018.24.6.560. PMID 30079951
- [Background] Sunuwar DR, Sangroula RK, Shakya NS, Yadav R, Chaudhary NK, Pradhan PMS. Effect of nutrition education on hemoglobin level in pregnant women: A quasi-experimental study. PLoS One. 2019 Mar 21;14(3):e0213982. doi: 10.1371/journal.pone.0213982. eCollection 2019. PMID 30897129
- [Derived] Rahman MJ, Rahman MM, Sarker MHR, Matsuyama R, Kakehashi M, Tsunematsu M, Ali M, Ahmed A, Hawlader MDH, Kawasaki H, Shimpuku Y. Impact of mobile health-based nutritional education on hemoglobin levels in anemic adolescent girls in rural Bangladesh: a randomized controlled trial. BMC Public Health. 2025 Jul 28;25(1):2567. doi: 10.1186/s12889-025-23687-z. PMID 40722070
- See also: Regional strategy for strengthening ehealth in the South-East Asia Region, WHO (2014-2020) — http://apps.who.int/iris/handle/10665/160760